CLINICAL TRIAL: NCT01823549
Title: Use of Nutritional Supplements and CAM (Complementary and Alternative Medicine) by Prostate and Breast Cancer Patients Undergoing Radiotherapy
Brief Title: Nutritional Supplements & Complementary/Alternative Medicine by Prostate & Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Steven Clinton, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-0240
Record Dates: First submitted 2013-03-28; First posted 2013-04-04 (Estimated); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer; Breast Cancer
Keywords: CAM; Alternative Medicine
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire administration — Ancillary studies

SUMMARY:
This study was a survey to determine the frequency of Complementary and Alternative Medicine (CAM) use in patients recently diagnosed with breast or prostate cancer who were starting radiation therapy. The survey was repeated at three time points to assess changes in CAM use over time.

ELIGIBILITY:
Inclusion/Exclusions

* Men that have histologically proven carcinoma of the prostate and have chosen some form of radiation therapy as their primary therapy for prostate cancer.
* Women who are undergoing external beam radiation therapy to the breast as primary or adjuvant therapy are eligible.
* All participants must be able to read and write.
* Subjects with dementia and mental retardation that complicates completing the questionnaires will not be enrolled.
* Subjects with known metastatic disease will be excluded.
* There are no age restrictions for this study.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men with clinically localized prostate cancer that have chosen external beam irradiation or brachytherapy or a combination for their treatment and women with localized breast cancer who are scheduled to begin external beam radiation therapy as a component of their primary or adjuvant therapy.
Sampling Method: Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2002-12-11 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Quantitate the various types of CAM therapy utilized by men with prostate cancer and women with breast cancer who are currently undergoing radiation. | Up to 1 year
  Quantitate the various types of CAM therapy utilized by men with prostate cancer and women with breast cancer who are currently undergoing radiation therapy at The James Cancer Hospital and Solove Research Institute. Nutrient supplements and alternative medication use is the primary focus of the assessment.
Determine if patients change their patterns of CAM use prior to, during, or after radiation treatment. | Up to 1 year
Assess quality of life using validated instruments during radiation therapy and determine if there is a correlation between CAM use and quality of life. | Up to 1 year
Assess radiation therapy toxicity using standardized criteria from the Oncology Nursing Society and determine if there is a correlation between CAM use and measures of toxicity. | Up to 1 year
To determine predictive factors for CAM and nutritional supplement use, such as age, race, income, education, marital status, or tobacco/alcohol use. | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Steven Clinton, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu